CLINICAL TRIAL: NCT07137130
Title: Development Of Adipose-Derived Mesenchymal Stem Cells Secretome (ADMSCS) Based Products From Stem Cell Conditioned Medium For Melasma Therapy
Brief Title: Secretome TGF Beta 3
Acronym: TGF Beta 3
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr.dr.Irma Bernadette, SpKK (K), Prof. M.D, Ph.D (Principal Investigator and Clinical Professor), Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TGF B3
Record Dates: First submitted 2025-08-06; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secretome raw material group (Experimental): Group A, the treatment group, used Secretome (raw material) 3ml Intradermal injection, Sunscreen in the morning and used Tretinoin cream 0,05% at night and cleanser which was used in the morning and evening before using the cream.
  Interventions: Drug: Concentrated secretome Injection 3 mL; Drug: Concentrated secretome Injection 3 mL with addition of TGF Beta 3
- Secretome raw material with addition of TGF Beta 3 group (Experimental): Group B, the treatment group, used Secretome (raw material) 3ml with addition of TGF Beta 3 Intradermal injection, Sunscreen in the morning and used Tretinoin cream 0,05% at night and cleanser which was used in the morning and evening before using the cream.
  Interventions: Drug: Concentrated secretome Injection 3 mL; Drug: Concentrated secretome Injection 3 mL with addition of TGF Beta 3

INTERVENTIONS:
Drug: Concentrated secretome Injection 3 mL — The secretome used in this research comes from mesenchymal stem cells from adipose tissue produced by Dr. Cipto Mangunkusumo Hospital Stem Cell Medical Technology. The secretome produced by mesenchymal stem cells is collected, centrifuged to separate it from debris, and followed by filtration with a 0.22 μm pore filter to ensure sterility. Next, the concentration process is carried out using tangential flow filtration with the Spin-X UF 500® concentrator, packaged, and stored at -80 degrees Celsius. The product used is a sterile product, which is tested for sterility and total protein content. When it is to be used, the secretome is removed from the freezer, warmed (thawing), and injected into the patient according to a predetermined method.
Drug: Concentrated secretome Injection 3 mL with addition of TGF Beta 3 — The secretome used in this research comes from mesenchymal stem cells from adipose tissue produced by Dr. Cipto Mangunkusumo Hospital Stem Cell Medical Technology. The secretome produced by mesenchymal stem cells is collected, centrifuged to separate it from debris, and followed by filtration with a 0.22 μm pore filter to ensure sterility. Next, the concentration process is carried out using tangential flow filtration with the Spin-X UF 500® concentrator, packaged, and stored at -80 degrees Celsius. The product used is a sterile product, which is tested for sterility and total protein content. When it is to be used, the secretome is removed from the freezer, warmed (thawing), and injected into the patient according to a predetermined method after the secretome is ready, TGF beta 3 will be added to secretome

SUMMARY:
A therapeutic modality currently being developed for melasma is secretome. Secretome is a bioactive molecule secreted by mesenchymal stem cells in a conditioned medium containing a large number of growth factors, cytokines, various macromolecules, and extracellular vesicles, including microvesicles and exosomes, that can stimulate various biological reactions, particularly in modulating new tissue formation. Secretome can provide a depigmenting effect by increasing the proliferation and migration of epidermal keratinocytes, which contain melanin pigment, in line with increased fibroblast synthesis.

Secretomes contain various cytokines and growth factors, one of which is transforming growth factor (TGF)-β. TGF-β is primarily secreted by fibroblasts (FB) and, to a lesser extent, by keratinocytes, and plays a crucial role in regulating melanocyte function. TGF-β has been reported to inhibit cAMP/protein kinase A signaling and induce GLI2, which then suppresses microphthalmia-associated transcription factor (MITF), a central transcription factor in melanogenesis. A study by Moon et al. in Korea examined TGF-β3. Moon et al. examined the effects of TGF-β3 on melanogenesis in human melanocytes co-cultured with skin cells irradiated with ultraviolet (UV) light, and in UV-irradiated human skin. The results showed that UVB irradiation or stem cell factor (SCF)/endothelin-1 (ET-1) increased melanogenesis. TGF-β3 effectively inhibited melanin accumulation and tyrosinase activity by downregulating the extracellular signal-regulated kinase (ERK)/microphthalmia-associated transcription factor (MITF) pathway. TGF-β3 increased the expression of keratinocyte differentiation markers.

Mechanistically, TGF-β3 inhibits melanogenesis by inhibiting MITF expression, which is regulated by ERK. TGF-β1 reduces MITF but at the risk of inducing skin fibrosis. However, in the study by Moon et al., the aforementioned TGF Beta 1 function was not found in TGF-β3. Furthermore, TGF-β3 restored skin differentiation function in UV-irradiated keratinocytes.

To date, there have been no clinical trials comparing intradermal injection of concentrated secretome with intradermal injection of concentrated secretome with the addition of TGF-β3 as a melasma therapy in Indonesia, thus encouraging researchers to conduct further research.

DETAILED DESCRIPTION:
Melasma is a pigmentation disorder in the form of brownish macules with irregular edges caused by dysfunctional melanogenesis. Melasma is more common in women with Fitzpatrick skin types IV-VI, namely those of Asian, Hispanic, and African descent, especially on sun-exposed areas of the face. Various epidemiological studies report that melasma can occur in all ethnicities, but the prevalence of melasma tends to be higher in East Asian (Japanese, Korean, and Chinese), Indian, Pakistani, Middle Eastern, and Mediterranean-African populations. In a 2014 study, melasma patients in Asia tended to be aged 21-64 years. The prevalence of melasma varies from place to place depending on race, skin phototype, and intensity of sun exposure. 4 Based on the distribution of lesions, melasma is clinically divided into 3 types: centrofacial (65%), malar (20%), and mandibular (15%).

Melasma is a disorder with multifactorial causes. Several trigger factors for melasma include genetic predisposition, exposure to ultraviolet (UV) light, hormonal influences, pregnancy, cosmetic use, consumption of photosensitizing medications, stress, and oxidative stress. One of the main triggering factors that can worsen melasma lesions is UV light.

Melasma impacts a person's appearance, causing psychosocial and emotional disturbances and a decreased quality of life. Generally, melasma patients often complain of embarrassment, low self-confidence, dissatisfaction, and a lack of desire to travel.According to the WHO, quality of life is an individual's perception of their position in life, both in the context of culture, value systems, goals, expectations, standards, and concerns. In 2003, Balkhrisnan et al. developed a Melasma Quality of Life Scale (MELASQoL) questionnaire consisting of 10 questions to assess the effects of melasma on emotional aspects, social relationships, and daily activities.12 The MELASQoL questionnaire contains questions covering 3 domains, namely emotional conditions (questions 1-4), social life (questions 5-7, and 10), and recreation (questions 8-9). A study by Aditya et al. has validated and assessed the reliability of the MELASQoL questionnaire prepared in Indonesian, namely MELASQoL-INA. The higher the MELASQoL score, the lower the person's quality of life.

Various treatment modalities are available for melasma, but none are satisfactory, and relapses often occur after therapy is discontinued.15,16 The mainstay of melasma therapy is sun avoidance and the use of broad-spectrum sunscreen. Other primary treatments for melasma include eliminating causative factors and using bleaching agents, such as hydroquinone (HQ). Hydroquinone at a concentration of 2-5% as a single therapy or in combination with tretinoin and topical corticosteroids (triple combination cream) is the gold standard for melasma therapy. However, this therapy has side effects if used long-term and without proper monitoring. Therefore, a more effective treatment modality is needed for melasma treatment.

Technological advances have resulted in the development of cosmeceutical products derived from natural and synthetic ingredients, some of which have been clinically and empirically tested and successfully commercialized. In Indonesia, the cosmetics industry market is growing relatively rapidly, with total cosmetic product sales in 2017 (Rp9.76 trillion) increasing by 12.9% compared to 2016 (Rp8 trillion), and cosmetic exports increasing by 20% with a transaction value of US$406 million. This indicates that researchers and developers in the cosmetics industry are continuously innovating to find new compound combinations or other modalities to support the growth of the cosmetics market.

One therapeutic modality currently being developed for melasma is secretome. Secretome is a bioactive molecule secreted by mesenchymal stem cells in a conditioned medium containing a large number of growth factors, cytokines, and various macromolecules, as well as extracellular vesicles, including microvesicles and exosomes, that can stimulate various biological reactions, particularly in modulating various new tissue formations. Secretome can provide a depigmenting effect by increasing the proliferation and migration of epidermal keratinocytes, which contain melanin pigment, in line with increased fibroblast synthesis.

Secretomes contain various cytokines and growth factors, one of which is transforming growth factor (TGF)-β. TGF-β is predominantly secreted by fibroblasts (FB) and to a lesser extent by keratinocytes and plays a crucial role in regulating melanocyte function. TGF-β has been reported to inhibit cAMP/protein kinase A signaling and induce GLI2, which in turn suppresses microphthalmia-associated transcription factor (MITF), a central transcription factor in melanogenesis. A study by Moon et al. in Korea examined TGF-β3. Moon et al. examined the effects of TGF-β3 on melanogenesis in human melanocytes co-cultured with skin cells irradiated with ultraviolet (UV) light, and in UV-irradiated human skin. The results showed that UVB irradiation or stem cell factor (SCF)/endothelin-1 (ET-1) increased melanogenesis. TGF-β3 effectively inhibited melanin accumulation and tyrosinase activity by downregulating the extracellular signal-regulated kinase (ERK)/microphthalmia-associated transcription factor (MITF) pathway. TGF-β3 increased the expression of keratinocyte differentiation markers.

Mechanistically, TGF-β3 inhibits melanogenesis by inhibiting MITF expression, which is regulated by ERK. 27,28 TGF-β1 reduces MITF but at the risk of inducing skin fibrosis. However, in the study by Moon et al., mentioned function of TGF Beta 1 was not found in TGF-β3. Furthermore, TGF-β3 restored skin differentiation function in UV-irradiated keratinocytes.

To date, no clinical trials have compared intradermal injection of concentrated secretome with intradermal injection of concentrated secretome with the addition of TGF-β3 as a melasma therapy in Indonesia, prompting researchers to conduct further research. The examination parameters include the mMASI score, mexameter score, dermoscopy, and Wood's lamp. Wood's lamp examination is used to help identify the location of melanin pigment in melasma lesions. Dermoscopy is a non-invasive examination to visualize subsurface structures that are invisible to the naked eye. Mexameter is a fast, easy, and accurate spectrometer measurement technique for measuring the melanin index and erythema index in skin based on light reflection and absorption. The mexameter examination functions to measure the severity of melasma objectively.33 The severity of melasma and evaluation of therapy response can be assessed subjectively using the mMASI score.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with melasma.
* Women without melasma and have areas of skin that are clinically free of lesions for SP control.
* 30-60 years old.
* Fitzpatrick skin type IV-V.
* Willing to be a research subject by signing a research consent form (Informed Consent).

Exclusion Criteria:

* Pregnant and breastfeeding women.
* Currently using hormonal contraception or have ever used contraception hormones in the last 6 months.
* Using topical therapy for melasma, for example corticosteroids, tretinoin, hydroquinone, and other therapies that whiten or brighten the skin in the last 2 weeks.
* Using topical triple combination cream therapy for at least 3 months and did not show significant improvement
* Using systemic therapy for melasma, for example antioxidants or tranexamic acid in the last 4 weeks.
* History of superficial peeling therapy in the last 4 weeks.
* History of deep peeling therapy, laser or mechanical abrasion in the last 6 months.
* Using drugs that are photosensitizers such as tetracycline, phenytoin, carbamazepine, spironolactone.
* History of blood clotting disorders or on blood thinning therapy.
* Allergy to tranexamic acid.
* Have other skin complaints that may interfere with the evaluation of melasma, for example post-inflammatory hyperpigmentation, Hori's nevus, Ota's nevus, pigmented contact dermatitis, and other pigmentation disorders
* Difficulty complying with treatment.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Estimated)
Dates: Start 2026-02-14 (Estimated); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change of Melasma Severity based on Patient's Tolerability Assesment (PtGA). | re-evaluation on day 14, 28, 42, 56 and day 84 of therapy
  one method of evaluating the response to therapy in melasma which is assessed subjectively by the patient. The response to therapy can be assessed as follows No or slight response: < 25% improvement Moderate response: 25% - 50% improvement Good response: 50% improvement - < 75% Excellent response: improvement > 75% The response is said to be good if the score is above 50% since the previous visit
Change of Melasma Severity based on modified Melasma Severity Index (mMASI) score | re-evaluation on day 14, 28, 42, 56 and day 84 of therapy
  The range of values for mMASI is between 0 and 24 which can then be divided into mild melasma (0-8), moderate (8-16), and severe (16-24). improvement occurs if the mMASI score decreases by <50% from the previous visit worsening if score persists or mMASI Score Increase >50% re-evaluation on day 14, 28, 42, 56 and day 84 of therapy
Change of Melasma Severity based on Dermoscopy | re-evaluation on day 84 of therapy
  based on Dermoscopy Telangiectasis score assessment using a 5-point dermoscopy-scale: 0 = No visible capillaries. 1 = Elongated capillaries accompanied by dilation, not visible to the naked eye. 2 = Moderate telangiectasis that is beginning to be visible to the naked eye. 3 = Severe telangiectasis characterized by reduced capillary loops. 4 = Very severe telangiectasis characterized by dilatation and loss of capillary loops.
Change of Melasma Severity based on Wood's Lamp | re-evaluation on day 84 of therapy
  Epidermal Type/ Dermal Typed/ Mixed Typed
Change of Melanin Index Based on Mexameter | re-evaluation on day 14, 28, 42, 56 and day 84 of therapy
  improves if there is a decrease in melanin levels > 50% from the initial visit It is said to be bad or persistent if there is no decrease in melanin levels or there is a decrease of <50%
Change of Erytema Index Based on Mexameter | re-evaluation on day 14, 28, 42, 56 and day 84 of therapy
  improves if there is a decrease in Erytema levels > 50% from the initial visit It is said to be bad or persistent if there is no decrease in erythema levels or there is a decrease of <50%

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Central Jakarta, D.k.i Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moon HR, Jung JM, Kim SY, Song Y, Chang SE. TGF-beta3 suppresses melanogenesis in human melanocytes cocultured with UV-irradiated neighboring cells and human skin. J Dermatol Sci. 2020 Aug;99(2):100-108. doi: 10.1016/j.jdermsci.2020.06.007. Epub 2020 Jun 24. PMID 32620316